CLINICAL TRIAL: NCT03671629
Title: Involving Clinical Pharmacists in Transitional Care to Reduce Drug-related Readmissions Among the Elderly - a Randomized Controlled Trial
Brief Title: Clinical Pharmacist Intervention to Reduce Drug-related Readmissions Among Older People
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Responsible Party: Principal Investigator, Maria Gustafsson, Principal Investigator, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UmU-2018-700
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Drug Use
Keywords: Clinical pharmacist; Elderly; Adherence; Drug-related readmission

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A group of physicians and clinical pharmacists will asses whether readmissions are drug-related or not. This group is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition to a standard medication review at the hospital, this group also receives an enhanced clinical pharmacist service during 180 days after discharge from the hospital.
  Interventions: Other: Enhanced clinical pharmacist service
- Control group (No Intervention): This group receives standard care, which might include a medication review at the hospital.

INTERVENTIONS:
Other: Enhanced clinical pharmacist service — The intervention includes regular medical chart reviews, multiple patient interviews and, if needed, collaboration with the primary care physician.
  Arms: Intervention group

SUMMARY:
This randomized controlled trial primarily investigates if a clinical pharmacist intervention can reduce drug-related readmissions among patients >75 years. The intervention targets the transfer between hospital and primary care. In brief, the intervention includes medical chart reviews and patient interviews during a period of 180 days.

DETAILED DESCRIPTION:
At discharge from the hospital, patients that meet the inclusion criteria are offered to participate in the study. At this point the investigators will also gather baseline data through questionnaires on self-reported adherence (MARS-5) and quality of life (EQ-5D). The participants are randomized to the different study arms according to a stratified procedure based on their cognitive function.

The intervention group will have their charts reviewed every second week and be contacted by the clinical pharmacist through phone within 7 and after 30 and 60 days respectively to discuss their medications. If possible drug-related problems are suspected during the interviews that cannot be solved immediately, the physician is contacted.

Both groups have a follow-up time of 30 and 180 days. After 30 and 180 days, the patients will once again report adherence and quality of life. All other data can be gathered from the medical charts.

ELIGIBILITY:
Inclusion Criteria:

* Living at home
* Acutely admitted
* Registered at one of ten pre-specified primary care health centers

Exclusion Criteria:

* Patients unable to communicate or who do not speak Swedish
* Patients scheduled for palliative care
* Patients admitted due to intoxication by alcohol or drug (non prescription)

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Time from discharge to first drug-related readmission | 180 days
  Survival analysis with drug-related readmission as endpoint

SECONDARY OUTCOMES:
Time from discharge to first drug-related readmission | 30 days
  Survival analysis with drug-related readmission as endpoint
Frequency of drug-related readmissions | 30 and 180 days
  Difference in total number of drug-related readmissions
Time from discharge to first drug-related readmission - subgroups with/without heart failure | 30 and 180 days
  Survival analysis among patients with/without heart failure
Time from discharge to first drug-related readmission - subgroups with/without cognitive impairment | 30 and 180 days
  Survival analysis among patients with/without cognitive impairment
Frequency of drug-related readmissions - subgroups with/without cognitive impairment | 30 and 180 days
  Subgroup analysis among patients with/without cognitive impairment
Frequency of drug-related readmissions - subgroups with/without heart failure | 30 and 180 days
  Subgroup analysis among patients with/without heart failure
Time from discharge to first all-cause hospital visit | 30 and 180 days
  Survival analysis with readmission or visit to the emergency department as endpoint
Frequency of all-cause hospital visits | 30 and 180 days
  Difference in total number of readmissions and visits to the emergency department
Self-reported adherence | 30 and 180 days
  Adherence to medications reported through MARS-5 ( Medication Adherence Rating Scale) and Swedish Prescribed Drug Register
Self assessed quality of life: EQ-5D-questionnaire | 30 and 180 days
  Health-related quality of life reported through the EQ-5D-questionnaire
Health economics | 180 days
  Cost for visits for (drug-related) readmissions and to visits to the Emergency Department compared between patients in the control group and intervention group.
Medication appropriateness | 180 days
  Medication appropriateness using the implicit Medication Appropriateness Index (MAI) and explicit tools in the form of the quality indicators published by the Swedish National Board of Health and Welfare and The European Union (EU)(7)-PIM list
Mortality | 30 and 180 days
  Survival analysis with death as endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gustafsson, Ph.D, Principal Investigator — Umeå University
Locations (1):
- Medical Centre, University Hospital of Umeå, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kindstedt J, Svahn S, Sjolander M, Glader EL, Lovheim H, Gustafsson M. Investigating the effect of clinical pharmacist intervention in transitions of care on drug-related hospital readmissions among the elderly: study protocol for a randomised controlled trial. BMJ Open. 2020 Apr 27;10(4):e036650. doi: 10.1136/bmjopen-2019-036650. PMID 32345700